CLINICAL TRIAL: NCT05477576
Title: Phase 1b/3 Global, Randomized, Controlled, Open-label Trial Comparing Treatment With RYZ101 to Standard of Care Therapy in Subjects With Inoperable, Advanced, SSTR+, Well-differentiated GEP-NETs That Have Progressed Following Prior 177Lu-SSA Therapy
Brief Title: Study of RYZ101 Compared With SOC in Pts w Inoperable SSTR+ Well-differentiated GEP-NET That Has Progressed Following 177Lu-SSA Therapy
Acronym: ACTION-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RayzeBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RYZ101-301
Record Dates: First submitted 2022-07-20; First posted 2022-07-28 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: GEP-NET; Gastroenteropancreatic Neuroendocrine Tumor; Gastroenteropancreatic Neuroendocrine Tumor Disease; Neuroendocrine Tumors; Carcinoid; Carcinoid Tumor; Pancreatic NET
Keywords: Neuroendocrine Tumors; SSTR+; GEP-NET; targeted radiotherapy; Gastroenteropancreatic Neuroendocrine Tumor; RayzeBio; Actinium; Ac 225; Dotatate; Everolimus; sunitinib; octreotide; lanreotide; PRRT; alpha emitter
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Neuroendocrine Tumors; Carcinoid Tumor; Adenoma, Islet Cell | interventions — Everolimus; Sunitinib; Octreotide; lanreotide

STUDY DESIGN:
Intervention Model Description: This study aims to determine the safety, pharmacokinetics (PK) and recommended Phase 3 dose (RP3D) of RYZ101 in Part 1, and the safety, efficacy, and PK of RYZ101 compared with investigator-selected standard of care (SoC) therapy in Part 2 in subjects with inoperable, advanced, well-differentiated, somatostatin receptor expressing (SSTR+) gastroenteropancreatic neuroendocrine tumors (GEP-NETs) that have progressed following treatment with Lutetium 177-labelled somatostatin analogue (177Lu-SSA) therapy, such as 177Lu-DOTATATE or 177Lu-DOTATOC (177Lu-DOTATATE/TOC), or 177Lu-high affinity [HA]-DOTATATE.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (4):
- Phase 1b - RYZ101 (Experimental): Part 1 is an uncontrolled dose de-escalation study to confirm the safety and determine the RP3D of RYZ101 based on Bayesian optimal interval design.
  Interventions: Drug: RYZ101
- Phase 3 - RYZ101 (Active Comparator): Actinium 225 radiolabeled somatostatin analog (SSA) for injection
  Interventions: Drug: RYZ101
- Phase 3 - Standard of Care (Active Comparator): Investigator's choice of standard of care between everolimus, sunitinib, octreotide, or lanreotide.
  Interventions: Drug: Everolimus; Drug: Sunitinib; Drug: Octreotide; Drug: Lanreotide
- Phase 3 - RYZ101, PK/ECG Substudy adhoc subcohort (Active Comparator): Actinium 225 radiolabeled somatostatin analog (SSA) for injection
  Interventions: Drug: RYZ101

INTERVENTIONS:
Drug: RYZ101 — RP3D as determined in Phase 1b
  Arms: Phase 1b - RYZ101; Phase 3 - RYZ101; Phase 3 - RYZ101, PK/ECG Substudy adhoc subcohort
Drug: Everolimus — Everolimus
  Arms: Phase 3 - Standard of Care
Drug: Sunitinib — Sunitinib
  Arms: Phase 3 - Standard of Care
Drug: Octreotide — High-dose octreotide
  Arms: Phase 3 - Standard of Care
Drug: Lanreotide — Lanreotide
  Arms: Phase 3 - Standard of Care

SUMMARY:
This study aims to determine the safety, pharmacokinetics (PK) and recommended Phase 3 dose (RP3D) of RYZ101 in Part 1, and the safety, efficacy, and PK of RYZ101 compared with investigator-selected standard of care (SoC) therapy in Part 2 in subjects with inoperable, advanced, well-differentiated, somatostatin receptor expressing (SSTR+) gastroenteropancreatic neuroendocrine tumors (GEP-NETs) that have progressed following treatment with Lutetium 177-labelled somatostatin analogue (177Lu-SSA) therapy, such as 177Lu-DOTATATE or 177Lu-DOTATOC (177Lu-DOTATATE/TOC), or 177Lu-high affinity [HA]-DOTATATE.

ELIGIBILITY:
Inclusion:

* Histologically proven, Grade 1-2 well differentiated, inoperable, advanced GEP-NETs (Ki67 ≤20%) Eastern Cooperative Oncology Group (ECOG) status 0-2. Ki67% <20% is not required for the ad hoc subcohort of the PK/ECG substudy.
* Progressive, SSTR-PET positive (i.e., Krenning score 3 or 4) GEP-NET (GI or pancreas) following 2-4 cycles of treatment with 177Lu-labeled SSA. Must have achieved disease control for at least 6 months following Lu-177 SSA (archival tissue is not required for the ad hoc subcohort of the PK/ECG substudy). No time limit is defined between 177Lu-SSA treatment and randomization. There must be at least 1 SSTR-PET imaging-positive measurable site of disease (according to RECIST v1.1) and no RECIST v1.1 measurable metastatic lesions that are SSTR imaging-negative.
* Adequate renal function, as evidenced by estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m2 (calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) (Levey et al. 2009)
* Adequate hematologic function, defined by the following laboratory results:
* Part 2: Hemoglobin concentration ≥5.0 mmol/L (≥8.0 g/dL); ANC ≥1000 cells/µL (≥1000 cells/mm3); platelets ≥75 x 109/L (75 x 103/mm3).
* Total bilirubin ≤3 x upper limit normal (ULN)
* Serum albumin ≥3.0 g/dL unless prothrombin time is within the normal range

Exclusion:

* Prior radioembolization
* Significant cardiovascular disease, such as New York Heart Association (NYHA) Class ≥II heart failure, left ventricular ejection fraction (LVEF) <40% or QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 ms for males and >470 ms for females.
* Resistant hypertension, defined as uncontrolled blood pressure (BP) >140/90 mmHg while on optimal doses of at least 3 antihypertensive medications with 1 being a diuretic (Whelton et al. 2018)
* Uncontrolled diabetes mellitus as defined by hemoglobin A1C (HgB A1C) ≥8%
* PRRT other than Lu-177 SSA (not applicable for ad hoc subcohort of the PK/ECG substudy)
* Any condition requiring systemic treatment with high-dose glucocorticoids within 14 days prior to first dose of study treatment and/or which cannot be stopped while on study. Inhaled or topical steroids are permitted.
* Prior history of liver cirrhosis or liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2022-03-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1b: RP3D | 56 days of study treatment
  Incidence of DLTs during the first 56 days of study treatment will be assessed.
Phase 3: PFS as determined by BICR | After the target number of 143 PFS events have occurred
  PFS will be defined as the time from the date of randomization until the date of progression (as determined by BICR from tumor assessments using RECIST v1.1) or death due to any cause, whichever occurs earlier.

CONTACTS AND LOCATIONS:
Overall Officials: Ye Yuan, MD, Study Director — RayzeBio Sr. Medical Director
Locations (52):
- United States (30):
  - Research Facility, Phoenix, Arizona
  - Research Facility, Duarte, California
  - Research Facility, Irvine, California
  - Research Facility, Los Angeles, California
  - Research Facility, Palo Alto, California
  - Research Facility, San Francisco, California
  - Research Facility, New Haven, Connecticut
  - Research Facility, Washington D.C., District of Columbia
  - Research Facility, Jacksonville, Florida
  - Research Facility, Miami, Florida
  - Research Facility, Tampa, Florida
  - Research Facility, Atlanta, Georgia
  - Research Facility, Iowa City, Iowa
  - Research Facility, Lexington, Kentucky
  - Research Facility, Glen Burnie, Maryland
  - Research Facility, Boston, Massachusetts
  - Research Facility, Troy, Michigan
  - Research Facility, Rochester, Minnesota
  - Research Facility, St Louis, Missouri
  - Research Facility, Omaha, Nebraska
  - Research Facility, New York, New York
  - Research Facility, Cleveland, Ohio
  - Research Facility, Columbus, Ohio
  - Research Facility, Portland, Oregon
  - Research Facility, Philadelphia, Pennsylvania
  - Research Facility, Pittsburgh, Pennsylvania
  - Research Facility, Nashville, Tennessee
  - Research Facility, Houston, Texas
  - Research Facility, Salt Lake City, Utah
  - Research Facility, Seattle, Washington
- Belgium (3):
  - Research Facility, Brussels
  - Research Facility, Leuven
  - Research Facility, Roeselare
- Brazil (3):
  - Research Facility, Brasília
  - Research Facility, Rio de Janeiro
  - Research Facility, São Paulo
- Canada (3):
  - Research Facility, London, Ontario
  - Research Facility, Toronto, Ontario
  - Research Facility, Montreal, Quebec
- France (6):
  - Research Facility, Clichy
  - Research Facility, Lille
  - Research Facility, Montpellier
  - Research Facility, Nantes
  - Research Facility, Vandœuvre-lès-Nancy
  - Research Facility, Villejuif
- Netherlands (3):
  - Research Facility, Amsterdam
  - Research Facility, Maastricht
  - Research Facility, Utrecht
- Research Facility, Seoul, South Korea
- Spain (3):
  - Research Facility, Barcelona
  - Research Facility, Madrid
  - Research Facility, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Taunk NK, Escorcia FE, Lewis JS, Bodei L. Radiopharmaceuticals for Cancer Diagnosis and Therapy: New Targets, New Therapies-Alpha-Emitters, Novel Targets. Cancer J. 2024 May-Jun 01;30(3):218-223. doi: 10.1097/PPO.0000000000000720. PMID 38753757